CLINICAL TRIAL: NCT02843347
Title: 1503 BMT CTN STRIDE Biorepository
Brief Title: STRIDE Biorepository
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, MD, Emory University
Other Study IDs: IRB00089102; 1U01HL128566 (NIH)
Record Dates: First submitted 2016-07-08; First posted 2016-07-25 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Anemia, Sickle Cell
Keywords: Biorepository; Genetics
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood will be collected, from participants who consent to the optional storage and future genetic testing of the sample provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biorepository substudy participants: Participants from the main study who give consent for the genetic testing substudy.
  Interventions: Procedure: Blood draw

INTERVENTIONS:
Procedure: Blood draw — Three tubes of blood (28.5 mL in total) will be obtained at the Baseline Visit. The sample will be stored for future research.

SUMMARY:
The STRIDE Biorepository is an optional substudy available to participants in "Bone Marrow Transplantation vs Standard of Care in Patients with Severe Sickle Cell Disease (BMT CTN 1503) (STRIDE)".

DETAILED DESCRIPTION:
A subset of sites for the main study "Bone Marrow Transplantation vs Standard of Care in Patients with Severe Sickle Cell Disease (BMT CTN 1503) (STRIDE)" (NCT02766465) will also participate in the biorepository portion of the study. The purpose of the biorepository is to examine DNA to learn if certain genes predict who will have serious complications of sickle cell disease. The STRIDE Biorepository is an optional substudy available to individuals enrolled in the main study, who are at a participating site. Participants in the main study who consent to take part in the biorepository will have blood drawn at the Baseline Visit. This blood will be shipped to Emory University in Atlanta Georgia and stored for future research.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 15 years old to less than 41 years old
* Severe sickle cell disease [any clinically significant sickle genotype, for example, Hemoglobin SS (Hb SS), Hemoglobin SC (Hb SC) or Hemoglobin SBeta thalassemia (Hb Sβ), or Hemoglobin S-OArab genotype] with at least 1 of the following manifestations:

  1. Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours;
  2. History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy);
  3. An average of three or more pain crises per year in the 2-year period preceding enrollment or referral (required intravenous pain management in the outpatient or inpatient hospital setting);
  4. Administration of regular red blood cell (RBC) transfusion therapy, defined as receiving 8 or more transfusions per year(in the 12 months before enrollment to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome);
  5. An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity ≥ 2.7 m/sec;
  6. Ongoing high impact chronic pain on a majority of days per month for at least 6 months.
* Adequate physical function as measured by all of the following:

  1. Karnofsky/Lansky performance score > or equal to 60
  2. Cardiac function: Left ventricular ejection fraction (LVEF) > 40%; or LV shortening fraction > 26% by cardiac echocardiogram or by Multi Gated Acquisition (MUGA) Scan
  3. Pulmonary function: Pulse oximetry with a baseline O2 saturation of ≥ 85% and diffusing capacity of the lung for carbon monoxide (DLCO) > 40% (corrected for hemoglobin)
  4. Renal function: Serum creatinine ≤ 1.5 x the upper limit of normal for age as per local laboratory and creatinine clearance >70 mL/min; or GFR > 70 mL/min/1.73 m2 by radionuclide Glomerular Filtration Rate (GFR)
  5. Hepatic function: Serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 times upper limit of normal as per local laboratory.

Exclusion Criteria:

* Human Leukocyte Antigen (HLA) typing prior to referral (consultation with hematopoietic cell transplantation (HCT) physician). However, if a subject has had HLA typing with accompanying documentation that relatives were not HLA typed and that a search of the unrelated donor registry was not performed the subject will be considered eligible. Documentation will be reviewed and adjudicated by the Protocol Officer or his/her designee.
* Uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment.
* Seropositivity for HIV
* Previous HCT or solid organ transplant
* Participation in a clinical trial in which the patient received an investigational drug or device must be discontinued at enrollment.
* A history of substance abuse as defined by version IV of the Diagnostic & Statistical Manual of Mental Disorders (DSM IV).
* Demonstrated lack of compliance with prior medical care (determined by referring physician).
* Pregnant or breast feeding females.
* Inability to receive HCT due to alloimmunization, defined as the inability to receive packed red blood cell (pRBC) transfusion therapy.

Additional Eligibility Criteria for Transplant after Biologic Assignment to the Donor Arm:

Participants assigned to the Donor Arm at the time of biologic assignment are subject to additional transplant eligibility criteria as specified below. Additional, repeat clinical assessments prior to transplant should be obtained in accordance with institutional policies and standards of care in the interest of good clinical practice.

* Participants must have liver magnetic resonance imaging (MRI) (at least 90 days prior to initiation of transplant conditioning) to document hepatic iron content is required for participants who are currently receiving ≥8 packed red blood cell transfusions for ≥1 year or have received ≥20 packed red blood cell transfusions (cumulative). Participants who have hepatic iron content ≥7 mg Fe/g liver dry weight by liver MRI must have a liver biopsy and histological examination/documentation of the absence of cirrhosis, bridging fibrosis, and active hepatitis (at least 90 days prior to initiation of transplant conditioning).
* Cerebral MRI/magnetic resonance angiogram (MRA) within 30 days prior to initiation of transplant conditioning. If there is clinical or radiologic evidence of a recent neurologic event (such as stroke or transient ischemic attack) subjects will be deferred for at least 6 months with repeat cerebral MRI/MRA to ensure stabilization of the neurologic event prior to proceeding to transplantation.
* Documentation of participant's willingness to use approved contraception method until discontinuation of all immunosuppressive medications. This is to be documented in the medical record corresponding with the consent conference.
* Have a suitably matched HLA donor
* Willing and able to donate bone marrow
* Absence of anti-donor HLA antibodies

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The biorepository will consist of research participants from the main study who consent to having extra blood drawn and stored for the purpose of future genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Genetic variants in persons with sickle cell disease | Baseline Visit
  A biorepository will be established for future genetic research of sickle cell disease. Blood samples will be drawn from participants at the Baseline Visit and will be stored until analyzed. Analysis will include learning more about the genetics behind complications of sickle cell disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University
Locations (40):
- United States (40):
  - Benioff Children's Hospital at Oakland, Oakland, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Gainsville, Gainesville, Florida
  - Foundation for Sickle Cell Research/Florida Sickle Inc., Hollywood, Florida
  - University of Miami, Miami, Florida
  - Grady Hospital, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Oschner Medical Center, New Orleans, Louisiana
  - Dana Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Dana Farber Cancer Institute/Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center/Albert Einstein School of Medicine, The Bronx, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Sciences Center, Houston, Texas
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - University of Texas/MD Anderson CRC, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia